CLINICAL TRIAL: NCT05339360
Title: Post-Market Clinical Follow-up Study on the ZNN™ Bactiguard ® Antegrade Femoral Nails (Implants and Instrumentation). A Multicenter, Prospective, Consecutive Series
Brief Title: ZNN Bactiguard Antegrade Femoral Nails PMCF Study
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2021-38T
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Femur Fracture; Osteotomy
Keywords: Intramedullary antegrade femoral nail; Bactiguard
MeSH Terms: conditions — Femoral Fractures | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ZNN Bactiguard Antegrade Femoral Nail: Subjects that have received or will receive the ZNN Bacitugard Antegrade Femoral Nail to treat femoral fractures or osteotomies according to the cleared/approved indications.
  Interventions: Procedure: Femoral fixation with intramedullary nails

INTERVENTIONS:
Procedure: Femoral fixation with intramedullary nails — Femoral fracture fixation Femoral Osteotomy

SUMMARY:
This is a multicenter, prospective, Post-market Clinical Follow-up (PMCF) Study on the ZNN Bactiguard Antegrade Femoral Nails. The objective of this study is to collect data confirming the safety, performance, and clinical benefit of the study device and instrumentation when used for the temporary internal fixation and stabilization of femoral fractures and osteotomies.

This is a CE-marked device already available on the market and the aim of the study is to comply with the post-market surveillance requirements.

DETAILED DESCRIPTION:
This study is a multicentre, prospective, post-market clinical follow-up study on the Zimmer Natural Nail (ZNN) Bactiguard Antegrade Femoral Nails.

The primary endpoint for this study is the assessment of performance by analyzing fracture healing within 12 months after fracture fixation. Fracture healing will be analyzed radiologically by the RUSH score adapted to the femur and clinically by the Fix-IT score.

The secondary endpoint is the assessment of safety, clinical benefit, and post-op fracture-related infection (FRI). Safety will be evaluated by recording and analyzing the incidence and frequency of complications and adverse events.

Relation of the events to implant, instrumentation and/or procedure should be specified. Clinical benefit will be assessed by recording patient-reported outcome measures (PROMs). FRIs will be classified according to the updated diagnostic algorithm defined by the FRI Consensus Group.

Data will be collected at 6 weeks, 3 months, 6 months and 1 year after fracture fixation.

The study will enroll patients implanted with the Zimmer Natural Nail Bactiguard Antegrade Femoral Nail according to the approved/cleared indications. The sample size for this study is 100 study cases, and up to 10 sites in EMEA will participate.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 or older
* Patient must have a signed EC-approved informed consent.
* Patient must have a femoral fracture (open, closed, monolateral, or bilateral) requiring surgical intervention or osteotomy and be eligible for fixation by intramedullary nailing. Patients with delayed treatment (initial treatment by external fixation due to swelling/ high energy trauma followed by definitive treatment by intramedullary nail) can also be included.
* Patient has been or is scheduled to be treated with the ZNN Bactiguard System Antegrade Femoral Nail
* Patient must be able and willing to complete the protocol required for follow-up
* Patients capable of understanding the surgeon's explanations and following his instructions

Exclusion Criteria:

Skeletally immature patients

* Medullary canal obliterated by a previous fracture or tumor
* Bone shaft having excessive bow or a deformity
* Lack of bone substance or bone quality, which makes stable seating of the implant impossible
* All concomitant diseases that can impair the operation, functioning or the success of the implant
* Insufficient blood circulation
* Infection
* Patient is unwilling to give consent.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, subjects with alcohol/drug addiction, known to be pregnant or breast feeding)
* Patient anticipated to be non-compliant and/or likely to have problems with maintaining follow-up program (e.g. patient with no fixed address, long-distance, plans to move during the course of study)
* Patients not expected to survive the duration of the follow-up program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of patients aged 18 or older with femur fractures or osteotomies implanted with the ZNN Bactiguard Antegrade Femoral Nail according to the approved/cleared indications.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Performance of the study device | 12 months after fracture fixation
  Analyzed as fracture healing 12 months after fracture fixation. Fracture healing will be analyzed radiographically and clinically. Radiographic healing is considered achieved when two or more cortices reach a score of two (2) on a version of the Radiographic Union-Scale in Tibial fractures (RUST) tool adapted for the femur, in A/P and lateral views. Clinical fracture healing will be assessed via the FiX-IT score.

SECONDARY OUTCOMES:
Safety assesment | 6 weeks and 3, 6, and 12 months after fracture fixation
  Recording and analyzing incidence and frequency of adverse events.
Oxford Hip Score | 3, 6, and 12 months after fracture fixation
  Patient-Reported Outcome Measures (PROMs) that documents hip function and pain. It's used as a surrogate to assess function and pain of the operated limb.
EQ-5D Health Questionnaire | 3, 6, and 12 months after fracture fixation
  Patient-reported outcome completed by the patient. It assesses the general health status of the patient and it can be used to derive a quality of life index used for health economics considerations.
Rate of fracture-related infections | 6 weeks and 3, 6, and 12 months after fracture fixation
  Fracture-related infections are diagnosed in accordance with the algorithm described in M McNally, G Govaert, M Dudareva, M Morgenstern, W J Metsemakers, EFORT Open Rev 2020;5:614-619.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (2):
- Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Santa Cruz de Tenerife, Spain
- Manchester Royal Infirmary, Manchester, Manchester, United Kingdom